CLINICAL TRIAL: NCT05236946
Title: Observation or Upfront Cranial RT in Oncogene Driver Mutated NSCLC With Asymptomatic Brain Metastases: A Phase III Randomized Controlled Trial
Brief Title: Observation or Upfront Cranial RT in Oncogene Mutated NSCLC With Asymptomatic BM: A Phase III RCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Anil Tibdewal, Dr. Anil Tibdewal, Associate Professor, Radiation Oncology, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRI/2020/08/027279; IEC/3470 (Other: Tata Memorial Hospital)
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Asymptomatic Brain Metastases; Driver Mutation Positive Non-small Cell Lung Cancer
Keywords: Asymptomatic brain metastases; EGFR mutation; Whole brain radiotherapy; Stereotactic radiosurgery; ALK rearrangement
MeSH Terms: interventions — Radiosurgery; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upfront Cranial Radiotherapy (Active Comparator): Stereotactic radiosurgery or Whole brain radiotherapy upfront in asymptomatic brain metastases
  Interventions: Radiation: Stereotactic radiosurgery/whole brain radiotherapy; Drug: Tyrosine kinase inhibitor
- Observation (Delayed Cranial Radiotherapy) (Experimental): Observation (Delayed Cranial radiotherapy) of Asymptomatic brain metastases
  Interventions: Drug: Tyrosine kinase inhibitor

INTERVENTIONS:
Radiation: Stereotactic radiosurgery/whole brain radiotherapy — SRS/ WBRT for asymptomatic brain metastases depending on the number of brain metastases
  Arms: Upfront Cranial Radiotherapy
Drug: Tyrosine kinase inhibitor — TKI

SUMMARY:
Tyrosine Kinase Inhibitors (TKIs) especially higher generation TKI have higher CNS penetration rates and have shown favorable response rates in brain metastases. Brain radiotherapy/surgery is the standard treatment in brain metastases especially symptomatic metastases, however, the role of local treatment especially in driver mutation-positive non-small cell lung cancer with asymptomatic brain metastases is being questioned given their potential side effects. No randomized trial has shown the superiority of early vs delayed cranial RT in asymptomatic BM of driver mutated NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with ECOG performance status of 0-2
3. Patients with pathologically proven diagnosis of NSCLC
4. Patients with positive oncogene mutation status (EGFR/ALK)
5. Patients with radiologically confirmed parenchymal brain metastases
6. Patients with asymptomatic Synchronous or Metachronous brain metastases
7. Patients willing for written informed consent and must be willing to comply with the specified follow-up schedule

Exclusion Criteria:

1. Patients with CSF dissemination only without any parenchymal brain metastases
2. Patients with brain metastases in the brain stem
3. Patients with prior history of radiation therapy to the brain
4. Patient not suitable for TKI therapy as per the medical oncologist
5. Pregnant or lactating females

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression free survival at 24 months | 2 year
  Intracranial progression free survival will be defined as the time from the date of randomization until the date of intracranial progression is documented. Death without intracranial progression will be considered as a competing event. Intracranial response will be graded as per the Response Assessment in Neuro-Oncology (RANO) guidelines for brain metastases

SECONDARY OUTCOMES:
Overall Survival | Upto 5-year
  Overall survival will be defined as the time from randomization until the date of death from any cause in the presence or absence of recurrence.
Progression free survival | upto 2 year
  Progression free survival will be defined from the date of randomization to the date of progression or the date of death whichever is earlier.
Neurocognition toxicity | Upto 12 months
  Neuro-cognition assessment will be done using HVLT-R (Total Recall) at baseline and at 3, 6 and 12 months for assessable patients
Toxicity using CTC v5.1 | Upto 2 years
  Toxicity assessment will be defined as per the common terminology criteria version 5.0 at baseline and at subsequent follow up till 2 years
Local Control | Upto 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
Protocol manuscript will be published and the results will be published in international peer-reviewed journal